CLINICAL TRIAL: NCT04334213
Title: A Randomized, Open-label, Multiple-dose, Crossover Clinical Trial to Investigate the Pharmacokinetic Drug Interactions and Safety After Oral Administration of D745, D150 and CKD-501 in Healthy Adults
Brief Title: A Clinical Trial to Investigate the Pharmacokinetic Drug Interaction and Safety of CKD-501, D745 and D150
Acronym: CKD-383
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A101_01DDI1927
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Period 1: CKD-501 - A single oral dose of 1 tablet under fasting conditions for 5 days.
  Period 2: CKD-501, D745, D150 - A single oral dose of 4 tablets under fasting conditions for 5 days (CKD-501: 1 tablet, D745: 1 tablet, D150: 2 tablets).
  Interventions: Drug: CKD-501; Drug: CKD-501, D745, D150
- Sequence 2 (Experimental): Period 1: CKD-501, D745, D150 - A single oral dose of 4 tablets under fasting conditions for 5 days (CKD-501: 1 tablet, D745: 1 tablet, D150: 2 tablets). Period 2: CKD-501 - A single oral dose of 1 tablet under fasting conditions for 5 days
  Interventions: Drug: CKD-501; Drug: CKD-501, D745, D150
- Sequence 3 (Experimental): Period 1: D745, D150 - A single oral dose of 3 tablets under fasting conditions for 5 days (D745: 1 tablet, D150: 2 tablets). Period 2: CKD-501, D745, D150 - A single oral dose of 4 tablets under fasting conditions for 5 days (CKD-501: 1 tablet, D745: 1 tablet, D150: 2 tablets).
  Interventions: Drug: D745, D150; Drug: CKD-501, D745, D150
- Sequence 4 (Experimental): Period 1: CKD-501, D745, D150 - A single oral dose of 4 tablets under fasting conditions for 5 days (CKD-501: 1 tablet, D745: 1 tablet, D150: 2 tablets). Period 2: D745, D150 - A single oral dose of 3 tablets under fasting conditions for 5 days (D745: 1 tablet, D150: 2 tablets).
  Interventions: Drug: D745, D150; Drug: CKD-501, D745, D150

INTERVENTIONS:
Drug: CKD-501 — QD, PO
  Arms: Sequence 1; Sequence 2
Drug: D745, D150 — QD, PO
  Arms: Sequence 3; Sequence 4
Drug: CKD-501, D745, D150 — QD, PO

SUMMARY:
A Clinical trial to investigate the pharmacokinetic drug interaction and safety of CKD-501, D745 and D150

DETAILED DESCRIPTION:
A Randomized, Open-label, Multiple-dose, Crossover Clinical Trial to Investigate the Pharmacokinetic Drug Interactions and Safety after Oral Administration of D745, D150 and CKD-501 in Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged between 19 and 55-year-old
2. Weight ≥ 55kg (men) or ≥ 50kg (women), with calculated body mass index(BMI) of 18.5 to 27.0 kg/m2
3. Women must meet one of the criteria written below:

   * Menopause (No menstruation for 2 years)
   * Sterilization (Hysterectomy or Oophorectomy, Tubal ligation etc.)
4. Men agree to contraception & won't donate sperm during the participation of clinical trial
5. Those who voluntarily decide to participate and agree to comply with the cautions after hearing and fully understanding the detailed description of this clinical trial

Exclusion Criteria:

1. Those who have clinically significant disease or medical history of Hepatopathy, Renal dysfunction, Neurological disorder, Immunity disorder, Respiratory disorder, Genitourinary system disorder, Digestive system disorder, Endocrine system disorder, Cardiovascular disorder, Blood tumor, Psychical disorder, Severe urinary tract infection
2. Those who have clinically significant dehydration or vulnerable to dehydration by poor oral intake
3. Those who receive intravenous administration of radioactive iodine contrast agents (for intravenous urography, venous cholangiography, angiography, computed tomography using contrast agents, etc.) within 48 hours before the first administration of investigational product
4. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
5. Those who have past medical history of gastrointestinal disorder (Crohn's disease, ulcerative colitis, etc. except simple appendectomy or hernia surgery), which affect the absorption of drug
6. Those who have history of hypersensitivity to active pharmaceutical ingredient (Lobeglitazone, Empagliflozin, Metformin) or additives.
7. Those who have the test results written below

   * AST, ALT > 1.25 times higher than upper normal level
   * Total bilirubin > 1.5 times higher than upper normal level
   * eGFR (estimated Glomerular Filtration Rate, which is calculated by MDRD) < 60 mL/min/1.73m2
   * "Positive" or "Reactive" test result of Hepatitis B & C, HIV, RPR
   * Under 5 min resting condition, systolic blood pressure >150 mmHg or <90 mmHg, diastolic blood pressure >100 mmHg or <50 mmHg
8. Those who have a drug abuse history within one year or positive reaction on urine drug screening test
9. Those who received following drugs, which may affect results of clinical trial and safety Ethical-the-counter (ETC) drugs and herbal medicines within 14 days before the first administration of the investigational drug Over-the-counter (OTC) drugs, health foods and vitamin preparations within 7 days before the first administration of the investigational product
10. Those who take barbiturate and related (causing induction or inhibition of metabolism) drug within 1 month before the first administration of investigational product
11. Those who exceeding an alcohol and smoke consumption criteria or can't stop smoking, consuming alcohol and caffeine during hospitalization period Criteria: Caffeine > 5 cups/day, Alcohol > 210 g/week, Smoke > 10 cigarettes/day
12. Those who took grapefruit before the first administration of investigational product or can't stop taking grapefruit during hospitalization period
13. Those who received investigational product by participating in other clinical trial within 6 months before the first administration of investigational product
14. Those who donated whole blood within 2 months or apheresis within 1 month
15. Those who received transfusion within 1 month
16. Those who are pregnant or breastfeeding
17. Those who are deemed inappropriate to participate in clinical trial by investigators

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of CKD-501, D745, D150 | Day 1, Day 3, Day 4 - Pre-dose (0 hour) / Day 5 - Pre-dose (0 hour), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours
  Cmax,ss: Maximum concentration of drug in plasma at steady state
AUCtau,ss of CKD-501, D745, D150 | Day 1, Day 3, Day 4 - Pre-dose (0 hour) / Day 5 - Pre-dose (0 hour), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours
  AUCtau,ss: Area under the plasma drug concentration-time curve within a dosing interval(τ) at steady state

SECONDARY OUTCOMES:
Cmin,ss of CKD-501, D745, D150 | Day 1, Day 3, Day 4 - Pre-dose (0 hour) / Day 5 - Pre-dose (0 hour), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours
  Cmin,ss: Minimum concentration of drug in plasma at steady state
Tmax,ss of CKD-501, D745, D150 | Day 1, Day 3, Day 4 - Pre-dose (0 hour) / Day 5 - Pre-dose (0 hour), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours
  Tmax,ss: Time to maximum plasma concentration at steady state
CLss/F of CKD-501, D745, D150 | Day 1, Day 3, Day 4 - Pre-dose (0 hour) / Day 5 - Pre-dose (0 hour), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours
  CLss/F: Apparent Clearance at steady state
Fluctuation of CKD-501, D745, D150 | Day 1, Day 3, Day 4 - Pre-dose (0 hour) / Day 5 - Pre-dose (0 hour), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours
  Fluctuation: Peak trough fluctuation within one dosing interval

CONTACTS AND LOCATIONS:
Overall Officials: Choon Ok Kim, M.D., PhD., Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Kim CO, Park H, Park MS, Kim D, Hong T, Shin Y, Jin BH. Evaluation of pharmacokinetic interactions between lobeglitazone, empagliflozin, and metformin in healthy subjects. Transl Clin Pharmacol. 2023 Mar;31(1):59-68. doi: 10.12793/tcp.2023.31.e4. Epub 2023 Mar 23. PMID 37034122